CLINICAL TRIAL: NCT07339592
Title: CHRONO-NUTRITION INTERVENTIONS FOR IMPROVING SLEEP QUALITY: The Impact of Last Meal Composition and Timing on Sleep Quality Among Medical Residents at Hospitals
Brief Title: This Trial Examines How Last Meal Composition and Timing Affect Sleep Quality and Circadian Gene Expression Among Medical Residents. Recruitment Not Yet Started; Study Begins Dec 2025 and Ends Dec 2026.
Acronym: CHRONO-MED
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Hadeel Ali Ghazzawi, Prof., University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: University of Jordan 491/2025
Record Dates: First submitted 2025-12-16; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Sleep Quality; Meal Timing; Circadian Rhythm; Medical Residents; Nutrition Intake
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Carbohydrate Last Meal (Experimental): Dinner ≈30% of daily kcal; ~80% of dinner kcal from carbs; consumed 3-4 h before sleep for 2 weeks.
  Interventions: Dietary Supplement: High-Carbohydrate Last Meal
- High-Protein Last Meal (Experimental): ≈30% of daily kcal; ~38-54% of dinner kcal from protein; consumed 3-4 h before sleep for 2 weeks.
  Interventions: Dietary Supplement: High-Protein Last Meal
- Balanced Standard last meal (Active Comparator): Standard balanced dinner (per usual guidelines), same timing (3-4 h pre-sleep) and 2 weeks duration.
  Interventions: Dietary Supplement: Balanced Standard Dinner

INTERVENTIONS:
Dietary Supplement: High-Carbohydrate Last Meal — Dinner ≈30% daily kcal; ~80% carb; taken 3-4 h before sleep for 2 weeks
  Arms: High-Carbohydrate Last Meal
Dietary Supplement: High-Protein Last Meal — Dinner ≈30% daily kcal; ~38-54% protein; 3-4 h before sleep for 2 weeks.
  Arms: High-Protein Last Meal
Dietary Supplement: Balanced Standard Dinner — Standard macronutrient distribution; same timing (3-4h pre-sleep) and 2-week duration.
  Arms: Balanced Standard last meal

SUMMARY:
This randomized controlled trial aims to evaluate the effects of last meal composition and timing on sleep quality and circadian gene expression among medical residents in Jordanian hospitals. Sleep disturbances are common in this population due to long working hours, high stress, and irregular eating schedules. Chrono-nutrition, the science of aligning food intake with circadian rhythms, may provide a practical approach to improving sleep and overall well-being.

Participants will be randomly assigned to one of three groups:

1. High-carbohydrate last meal (≈80% of dinner calories from carbohydrates),
2. High-protein last meal (≈40-50% of dinner calories from protein),
3. Control group consuming a balanced standard meal. Each participant will consume the assigned meal 3-4 hours before bedtime for two weeks. Sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI) and smartwatch-derived parameters, while salivary samples collected pre- and post-intervention will be analyzed for CLOCK and BMAL1 gene expression. The study will also include dietary, anthropometric, and physical activity assessments.

This study has been approved by the Institutional Review Board of the University of Jordan (IRB No. 491/2025). Recruitment has not yet started. Enrollment is expected to begin in December 2025, with primary data collection completed by June 2026 and final study completion by December 2026.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled and working in Jordanian hospitals.
* Not currently following a specific diet or weight-loss program.
* Willing to comply with study protocol and intervention meals for two weeks. Provide written informed consent before participation.

Exclusion Criteria:

* Presence of any chronic medical condition (e.g., diabetes, thyroid disorders, gastrointestinal, cardiovascular, or respiratory diseases).
* Diagnosed sleep disorders, such as insomnia, sleep apnea, or restless legs syndrome.
* Mental health disorders (stress, anxiety, or depression diagnosed or medicated).
* Pregnancy or lactation.
* Use of medications or herbal supplements known to affect sleep (e.g., melatonin, chamomile, ashwagandha, lavender).
* Caffeine dependence exceeding moderate levels ( >400 mg caffeine/day).

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Sleep Quality (PSQI Global Score) | Baseline and 2 weeks post-intervention
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI) before and after the 2-week intervention. The PSQI total score (0-21) will quantify subjective sleep quality; higher scores indicate poorer sleep

SECONDARY OUTCOMES:
Change in CLOCK Gene Expression | Baseline and 2 weeks post-intervention
  CLOCK mRNA expression will be measured in salivary samples collected pre- and post-intervention using RT-PCR. Relative quantification (ΔCt method) will determine expression changes.
Change in BMAL-1 Gene Expression | Baseline and 2 weeks post-intervention
  BMAL-1 mRNA levels will be analyzed in the same saliva samples via real-time PCR. Changes will be compared across meal groups.
Change in Total Sleep Duration | 1 week baseline and 2 weeks during intervention
  Total sleep duration will be objectively measured using smartwatch data and expressed as average nightly sleep duration.
  Unit of Measure: Minutes per night
Change in Sleep Efficiency | 1 week baseline and 2 weeks during intervention
  Sleep efficiency will be calculated as the percentage of total sleep time divided by time in bed using smartwatch data.
  Unit of Measure: Percentage (%)
Change in Sleep Stage Distribution | 1 week baseline and 2 weeks during intervention
  Sleep stage distribution (light, deep, and REM sleep) will be assessed using smartwatch data and expressed as percentage of total sleep time.
  Unit of Measure: Percentage (%)
Change in Average Heart Rate During Sleep | 1 week baseline and 2 weeks during intervention
  Average heart rate during sleep will be measured using smartwatch data. Unit of Measure: Beats per minute (bpm)

CONTACTS AND LOCATIONS:
Overall Officials: Hadeel A Ghazzawi, professor, Principal Investigator — The University of Jordan School of Agriculture
Locations (1):
- University of Jordan Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No